CLINICAL TRIAL: NCT00171548
Title: Project to Promote the Evaluation of Cardiovascular Risk in Clinical Practice, and Assess Its Evolution After the Implementation of Multifactorial Preventive Strategy Aimed at Reducing the Level of Global Risk (SCORE Algorithm) in Subjects With Metabolic Syndrome and a Risk Level of 5%
Brief Title: Cardiovascular Risk Evaluation in Clinical Practice in Metabolic Syndrome Patients
Status: Completed | Type: Observational
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis
Other Study IDs: CVAL489AIT05
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2008-09-22 (Estimated); Status verified 2008-09

CONDITIONS: Metabolic Syndrome
Keywords: Metabolic syndrome, cardiovascular risk reduction
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Metabolic syndrome is commonly defined as a set of risk factors and abnormalities that markedly increase the risk of cardiovascular events. Its relevance has been confirmed by a recent population-based survey of subjects aged 40-79 years indicating that the prevalence of metabolic syndrome in Italy is 34.1% if diagnosed using WHO criteria and 17.8% if diagnosed using the NCEP-ATPIII criteria.

On the basis of the above considerations, the aim of this study is to promote the use of the SCORE algorithm for estimating cardiovascular risk, and to evaluate its evolution in patients with metabolic syndrome after the implementation of a multifactorial preventive strategy, with particular reference to the correction of lifestyle, hypertension and dyslipidemia.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both genders aged 40-65 years.
* A diagnosis of metabolic syndrome formulated on the basis of the criteria proposed by the NCEP - Adult Panel III: i.e. the presence of at least three of the following conditions:

  1. Waist circumference >102 cm in men and >88 cm in women
  2. Triglyceridemia 150 mg/dl
  3. HDL cholesterol <40 mg/dl in men and <50 mg/dl in women
  4. Sitting arterial pressure 130/85 mmHg
  5. Fasting glycemia 110 mg/dl
* A risk of cardiovascular death of >5% at the current age of the patient or >5% if projected to an age of 60 years, as calculated by means of the SCORE algorithm using the table based on the total/HDL cholesterol ratio relating to low-risk populations and appropriate for Italy.
* Written informed consent.

Exclusion Criteria:

* Women who have not been in menopause for at least one year or are not surgically sterile, and do not use an effective contraceptive method, such as spermicidal barrier methods or intrauterine devices. The use of oral contraceptives is not allowed.
* Known or suspected hypersensitivity to valsartan and/or fluvastatin, or other contraindications to their use;
* A positive history of ischemic heart disease, peripheral artery disease or cerebral vasculopathy;
* Patients with an SBP of 180 mmHg and/or DBP of 110 mmHg.
* Patients with severe medical conditions which, in the judgement of the Investigator, contraindicate trial participation or significantly limit life expectancy;
* Treatment with drugs able to modify the lipid profile (ongoing or in the three months preceding trial entry);
* Patients unable to follow the planned protocol procedures or sign the informed consent form.

Ages: 40 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2004-10; Primary Completion 2007-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Pharmaceuticals, Basel, Switzerland